CLINICAL TRIAL: NCT05156502
Title: An Open-Label, Interventional, Controlled Study To Assess The Performance And Tolerance Of Pixel CO2-Alma Fractionated Laser in Women Affected by GenitoUrinary Syndrome of Menopause (GSM)
Brief Title: To Assess Signs and Symptoms in Women Affected by GSM After One Cycle of Pixel CO2-Alma Fractionated Laser
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. Filippo Murina (Other)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor-Investigator, Dr. Filippo Murina, Responsabile Servizio di Patologia del tratto genitale inferiore, ASST Fatebenefratelli Sacco
Organization: ASST Fatebenefratelli Sacco (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSSM-2020-03.1
Record Dates: First submitted 2021-10-27; First posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Genitourinary Syndrome of Menopause (GSM); Vaginal Dryness; Burning; Pain; Dyspareunia; Dysuria
Keywords: Genitourinary syndrome of menopause (GSM); Fractionated Laser; Vaginal dryness.; dyspareunia
MeSH Terms: conditions — Paresthesia; Pain; Dyspareunia; Dysuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fractionated Laser (Experimental)
  Interventions: Device: Fractionated Laser (Pixel CO2-Alma)
- Fractionated.Laser (Active Comparator)
  Interventions: Device: Fractionated Laser (Pixel CO.2-Alma)

INTERVENTIONS:
Device: Fractionated Laser (Pixel CO2-Alma) — The Laser will be administered at baseline (visit 2, day 0), at visit 3 (day 28) and at visit 4 (day 56) into vagina and vestibule, following the IFU of the device.
  Arms: Fractionated Laser
Device: Fractionated Laser (Pixel CO.2-Alma) — Device: Fractionated Laser (Pixel CO2-Alma) The Laser will be administered at baseline (visit 2, day 0), at visit 3 (day 28) and at visit 4 (day 56) into vagina only, following the IFU of the device.
  Arms: Fractionated.Laser

SUMMARY:
Genitourinary syndrome of menopause (GSM) occurs in approximately 50% of menopausal women but is both underrecognized and undertreated despite numerous treatment options. Vaginal dryness, irritation, dyspareunia, urinary frequency, and urinary urgency are some of the more common symptoms that can have a negative effect on women's lives and relationships. In particular, dyspareunia is localized in the vestibule with specific trophic changes more evident than those localized in vagina. The CO2 fractionated laser, has also been found to be useful in several studies for the treatment of vaginal atrophy.

In this open comparative study, 70 female menopausal subjects aged between 40 and 70 years old at inclusion, having symptoms of GSM (Vaginal dryness, burning/pain, dyspareunia,dysuria), have given her informed consent and meet all the eligibility criteria, will be enrolled. The two groups of comparison will be 35 subjects treated into vagina and vestibule, versus 35 subjects treated into vagina, only. Subjects will come to a total of 6 visits over a period of 3 months.

The primary objective of the study is to evaluate the performance and safety of Pixel CO2-Alma Fractionated Laser comparing its administration into vagina and vestibule versus into vagina, only. The evaluated outcomes are vaginal dryness, burning/pain, dyspareunia, sensitivity to touch at Swab test, Female Sexual Function Index (FSFI) and Vulval Pain Functional Questionnaire (VQ) at day 84 and 120 and the safety during all the study. The secondary objectives are the evaluation of vaginal and vestibular trophism, measured by Vaginal Health Index (VHI) and Vestibular Health Score (VHS) at the FU visits.

ELIGIBILITY:
Inclusion Criteria:

* menopausal women aged between 40 and 70 years old (defined as Absence of menstruation for 12 consecutive months).
* women affected by Genitourinary syndrome of menopause (GSM) with Vaginal dryness, burning/pain, dyspareunia, dysuria.
* women not treated with Replacement therapy with estrogen and progestogen (HT) or estrogen alone (ET) or selective estrogen receptor modulators (SERMS) in the last 3 months

Exclusion Criteria:

* hypersensitivity to laser
* clinically significant findings on physical examination
* any chronic medical condition or psychologic disorder that per opinion of the Principal Investigator would make the patient ineligible for the study
* vulvo-vestibular lesion not related with GSM
* active vaginal or vulvar infections (e.g., herpes, candida, STIs)
* prolapse beyond the hymen
* subject has a history of scarring alteration (ie, keloid formation)
* unknown past or active history of vaginal bleeding disorders
* any condition or behavior indicating to the Principal Investigator that the Subject is unlikely to be compliant with study procedures and visits

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women affected by Genitourinary syndrome of menopause (GSM) with Vaginal dryness, burning/pain, dyspareunia, dysuria
Enrollment: 70 (Estimated)
Dates: Start 2022-01-30 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Vaginal dryness by Visual Analogue Scale | 120 days
  The changing will be measured by Visual Analogue Scale (VAS) mean values from baseline to day 84 (visit 5), and 120 (final visit) in each group separately and in the two groups in comparison. The minimum score is 0 and the maximum score is 10, where 0 represents no symptoms and 10 represents severe symptoms
Burning/pain by Visual Analogue Scale | 120 days
  The changing will be measured by Visual Analogue Scale (VAS) mean values from baseline to day 84 (visit 5), and 120 (final visit) in each group separately and in the two groups in comparison. The minimum score is 0 and the maximum score is 10, where 0 represents no symptoms and 10 represents severe symptoms
Dyspareunia by Visual Analogue Scale | 120 days
  The changing will be measured by Visual Analogue Scale (VAS) mean values from baseline to day 84 (visit 5), and 120 (final visit) in each group separately and in the two groups in comparison. The minimum score is 0 and the maximum score is 10, where 0 represents no symptoms and 10 represents severe symptoms
Pain/sensitivity to touch at Swab test by Visual Analogue Scale. | 120 days
  The changing will be measured by Visual Analogue Scale (VAS) mean values from baseline to day 84 (visit 5), and 120 (final visit) in each group separately and in the two groups in comparison. The minimum score is 0 and the maximum score is 10, where 0 represents no symptoms and 10 represents severe symptoms
Sexual Function by Female Sexual Function Index | 120 days
  Sexual function will be evaluated at baseline and after 84 and 120 days by the Italian validated translation of the Female Sexual Function Index (FSFI), a self-report instrument consisting of 19 items that assess sexual function over the past 4 weeks in six areas: sexual desire, arousal, lubrication, orgasm, satisfaction, and pain. Mean value in each group separately and in the two groups in comparison will be analyzed.
Vulval Pain by Vulval Pain Functional Questionnaire | 120 days
  The Vulval Pain Functional Questionnaire (VQ) will be used to quantify the extent that pelvic pain is affecting the patients. A numerical value is assigned to each response. The higher the score the greater the functional limitation. A diminishing score represents improvement.
Incidence of Treatment-Emergent Adverse Events/ Adverse Device Events/ Serious Adverse Events/ Serious Adverse Device Events [Safety and Tolerability] | up to 120 days
  The incidence will be calculated by searching for Adverse Event (AE), Adverse Device Event ADE, Serious Adverse Event (SAE), Serious Adverse Device Event (SADE) at each visit

SECONDARY OUTCOMES:
Vestibular Trophism by Vaginal Health Index | 120 days
  The changing from baseline to day 84 (visit 5) and 120 (final visit) for Vaginal Health Index (VHI) mean value in each group separately and the changing in Arm A in comparison with that occurred in Arm B. The VHI score evaluates 5 parameters (vaginal elasticity, vaginal secretions, vaginal pH, epithelial mucous membrane, vaginal hydration) and to obtain a final score defining the degree of atrophy in the genitourinary tract by assigning a single score to each parameter. The minim score is 5 and the maxim is 25.
Vestibular Trophism by Vestibular Health Score | 120 days
  Vestibular Health Score (VHS) will be used by the Investigator evaluating 5 parameters (Petechiae, Pallor, Fragility, dryness, Erythema) and to obtain a final score defining the degree of atrophy. Each item is scored on a Likert scale between 0 =absent and 3 =severe. Total scores range from 0 to 15.

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale dei Bambini V Buzzi, Milan, Italy